CLINICAL TRIAL: NCT06654752
Title: Streamlined Treatment of Pulmonary Exacerbations in Pediatrics Randomized Controlled Trial (STOP PEDS RCT)
Brief Title: Streamlined Treatment of Pulmonary Exacerbations in Pediatrics
Acronym: STOP PEDS RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington, the Collaborative Health Studies Coordinating Center (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOP PEDS RCT
Record Dates: First submitted 2024-10-14; First posted 2024-10-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; oral antibiotics; pulmonary exacerbation; pediatric
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Antibiotics (Experimental): Increased airway clearance plus early initiation of oral antibiotics
  Interventions: Other: Immediate Oral Antibiotics
- Tailored Therapy (Experimental): Increased airway clearance alone, with addition of oral antibiotics for worsening symptoms or failure to improve
  Interventions: Other: Tailored Treatment: Oral Antibiotics only if Additional Treatment needed

INTERVENTIONS:
Other: Immediate Oral Antibiotics — Increase airway clearance and start 14 days of preselected oral antibiotics right away
  Arms: Immediate Antibiotics
Other: Tailored Treatment: Oral Antibiotics only if Additional Treatment needed — Increase airway clearance and start preselected oral antibiotics later if symptoms get worse or do not get better according to prespecified criteria
  Arms: Tailored Therapy

SUMMARY:
The STOP PEDS RCT is a multicenter, parallel, open label randomized controlled trial evaluating the long-term (one year) and short-term safety and efficacy of two antibiotic treatment strategies for the management of outpatient pulmonary exacerbations (PEx) in the pediatric CF population.

DETAILED DESCRIPTION:
The STOP PEDS pilot study demonstrated that a randomized trial of treatment strategies for mild pulmonary exacerbations (PEx) in children with CF was feasible and that assignment to a tailored therapy arm (defined below) may reduce antibiotic exposure.

Based on the research priorities identified by CF families and clinicians and the results of the pilot study, the STOP PEDS RCT is a multicenter, parallel, open label randomized controlled trial evaluating the long-term (one year) and short-term safety and efficacy of two antibiotic treatment strategies for the management of outpatient PEx in the pediatric CF population. The two treatment arms are immediate antibiotics and tailored therapy. In both arms, participants will be instructed to increase airway clearance at the onset of an eligible PEx. In the immediate antibiotics arm, they will also begin 14 days of oral antibiotics preselected by their primary CF providers, while in the tailored therapy they will only begin antibiotics if prespecified criteria for worsening symptoms or failure to improve are met.

The STOP PEDS study will enroll three cohorts. In the main cohort, children ages 6-18 on highly effective modulator therapy (HEMT) will be enrolled when well and followed for 12 months. Participants will be randomly assigned to a treatment arm and maintain that treatment assignment for all subsequent eligible PEx during their 12-month enrollment period. Two additional pilot cohorts, the preschool cohort (children ages 3 to 5 on HEMT) and the non-HEMT cohort (children ages 6-18 not eligible for HEMT), will be enrolled in parallel pilot studies. Participants will enroll when well and be followed through one randomized PEx.

Participants in the STOP PEDS RCT at selected sites will have the opportunity to enroll in optional substudies if eligible. These substudies include:

* Clinic throat swab substudy
* Home throat and nasal swab substudy
* Remote monitoring substudy (Home monitoring of lung function, vital signs, activity and sleep)

ELIGIBILITY:
Inclusion Criteria:

1. Age

   1. For main cohort and non-HEMT cohort: age 6 to <19 years
   2. For preschool cohort: age 3 to <6 years
2. Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype and one or more of the following criteria:

   1. sweat chloride ≥ 60 mEq/liter
   2. two disease-causing variants in the cystic fibrosis transmembrane conductive regulator (CFTR) gene
3. Written informed consent (and assent when applicable) obtained from participant or participant's legal representative and ability of participant to comply with the requirements of the study
4. Highly Effective Modulator Therapy

   1. For main cohort and preschool cohort: Taking ETI or ivacaftor for at least 3 months at enrollment
   2. For non-HEMT cohort: not eligible for HEMT based on CFTR genotype or eligible but not taking for at least 3 months and no plans to start HEMT in the next year, and also not taking tezacaftor-ivacaftor or lumacaftor-ivacaftor for at least 3 months
5. For main cohort and non-HEMT cohort: able to perform acceptable and reproducible spirometry
6. For main cohort and non-HEMT cohort: ppFEV1 ≥ 50% predicted at enrollment based on the Global lung Initiative (GLI) reference equations
7. Ability to receive text messages and access the internet

Exclusion Criteria:

1. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the individual or the quality of the data
2. Receiving an acute course of oral or IV antibiotics at the time of enrollment or within the 14 days prior to enrollment. Individuals may be re-screened ≥21 days after completion of antibiotics if they are at their baseline state of health, per self-report
3. Treatment with systemic corticosteroids at enrollment or within the 14 days prior to enrollment. Individuals may be re- screened ≥21 days after completion of systemic corticosteroids if they are at their clinical baseline, per self-report
4. History of solid organ transplant
5. History of positive culture for Mycobacterium abscessus in the 12 months prior to enrollment
6. Treatment with antibiotics for any non-tuberculous mycobacteria (NTM) at enrollment
7. Three or more IV antibiotic-treated PEx in the 12 months prior to enrollment
8. Treatment with chronic oral antibiotics other than azithromycin at enrollment
9. Treatment with systemic corticosteroids for allergic bronchopulmonary aspergillosis (ABPA) in the 12 months prior to enrollment

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 430 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
One-year change in pulmonary function by spirometry-measured ppFEV1 | 1 year
  Compare the difference in pulmonary function between arms by evaluating change in spirometry-measured percent predicted forced expiratory volume (ppFEV1). A spirometry test measures the amount of air a person can forcibly exhale after a deep breath (forced vital capacity, or FVC) and the amount of air they can exhale in one second (forced expiratory volume in one second, or FEV1). A lower measured value compared to the reference value indicates lung disease.

SECONDARY OUTCOMES:
One-Year change in pulmonary function by LCI | 1 year
  Compare the difference in pulmonary function between arms by evaluating change in Lung Clearance Index (LCI). LCI increases when there is lung disease, which causes ventilation inhomogeneity. LCI is calculated as the number of lung volume turnovers (cumulative expired volume divided by the functional residual capacity [FRC]) required to reduce end-tidal nitrogen concentration to 1/40th of the original level.

OTHER OUTCOMES:
Recovery to baseline by ppFEV1 and CRISS following a PEx | 28 days
  Compare recovery to baseline between arms over the 28-day period after the first pulmonary exacerbation (PEx), by spirometry-measured percent predicted forced expiratory volume (ppFEV1), and after all pulmonary exacerbations, measured by CRISS symptom scores. The Chronic Respiratory Infection Symptom Score (CRISS) ranges from 0 to 100, with higher scores indicating more symptoms.
Recovery to baseline by Lung Clearance Index (LCI) | 28 days
  Compare recovery to baseline between arms over the 28-day period after the first pulmonary exacerbation (PEx) in LCI, and after all exacerbations for symptom scores. The Chronic Respiratory Infection Symptom Score (CRISS) ranges from 0 to 100, with higher scores indicating more symptoms.
Safety Endpoint 1: Cumulative oral antibiotic exposure | 1 year
  Compare cumulative oral antibiotic exposure in each treatment arm.
Safety Endpoint 2: Number of respiratory illnesses | 1 year
  Compare the number of respiratory illnesses reported over the study period in each treatment arm.
Safety Endpoint 3: Proportion of respiratory illnesses treated with antibiotics during PEx | 28 days
  Compare the proportion of respiratory illnesses treated with antibiotics during the 28-day pulmonary exacerbation (PEx) treatment period in each treatment arm.
Safety Endpoint 4: Number of PEx treated with IV antibiotics | 1 year
  Compare the number of pulmonary exacerbations (PEx) treated with IV antibiotics over the study period in each treatment arm.
Safety Endpoint 5: Proportion of PEx failing to recover to baseline symptoms at Day 28 | 28 days
  Compare the proportion of pulmonary exacerbations (PEx) failing to recover to baseline symptoms at Day 28 in each treatment arm.
Safety Endpoint 6: Proportion of PEx with ppFEV1 below baseline at Day 28 | 1 year
  Compare the proportion of pulmonary exacerbations (PEx) with spirometry-measured percent predicted forced expiratory volume (ppFEV1) below baseline at Day 28 in each treatment arm.
Safety Endpoint 7: Time from initial randomized PEx to next respiratory illness | 1 year
  Compare the time from initial randomized pulmonary exacerbation (PEx) to next respiratory illness in each treatment arm.
Safety Endpoint 8: Targeted adverse events (patient report of antibiotic side effects during PEx) | 1 year
  Compare the targeted adverse events (patient report of antibiotic side effects during pulmonary exacerbation period) in each treatment arm.
Safety Endpoint 9: Treatment-emergent CF microorganisms on clinical respiratory cultures | 1 year
  Compare treatment-emergent CF microorganisms on clinical respiratory cultures in each treatment arm.
Qualitative Assessment 1: Caregivers' experience managing study treatment | 1 year
  To understand benefits and challenges associated with assigned treatment through targeted qualitative interviews of caregivers we will describe caregivers' experience managing study treatment and report themes that emerge regarding caregivers' experiences.
Qualitative Assessment 2: Study treatment impact on child and family daily life | 1 year
  To understand benefits and challenges associated with assigned treatment through targeted qualitative interviews of caregivers we will evaluate study treatment impact on child and family daily life and report themes that emerge regarding caregivers' experiences.
Health care costs 1: Total estimated cost of antibiotics | 1 year
  Compare total estimated cost of antibiotics used over the course of the study between treatment arms.
Health care costs 2: Health care utilization | 1 year
  Compare health care utilization over the course of the study between treatment arms, including number of primary care visits and number of emergency room visits.
Health care costs 3: Parent work productivity measures (WPAI) | 1 year
  To compare parent Work Productivity and Activity Impairment (WPAI) measures between study arms. The WPAI includes four scores assessing absenteeism, presenteeism, work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment in the last seven days. Scores range from 0 to 100, with higher scores indicating greater impairment.
Preschool and non-HEMT Pilot Cohort Primary Feasibility | 28 days
  Estimate the proportion of preschool and non-HEMT (Highly Effective Modulator Therapy) participants randomized to the tailored therapy arm that has no antibiotic exposure in the 28 days following a pulmonary exacerbation (PEx).
Preschool and non-HEMT Pilot Cohort Safety Endpoint 1: ppFEV1 and LCI recovery | 28 days
  Compare percent predicted forced expiratory volume (ppFEV1) and Lung Clearance Index (LCI) recovery using Day 28 values compared to nearest pre-PEx baseline measure in both treatment arms.
Preschool and non-HEMT Pilot Cohort Safety Endpoint 2: Time to symptom recovery | 28 days
  Compare time to symptom recovery (number of days to recover to baseline CRISS score) between treatment arms. The Chronic Respiratory Infection Symptom Score (CRISS) ranges from 0 to 100, with higher scores indicating more symptoms.
Preschool and non-HEMT Pilot Cohort Safety Endpoint 3: Targeted adverse events | 28 days
  Compare targeted adverse events (participant report of antibiotic side effects during PEx period) between treatment arms.
Preschool and non-HEMT Pilot Cohort Safety Endpoint 4: Treatment-emergent CF microorganisms | 28 days
  Compare treatment-emergent CF microorganisms on clinical respiratory cultures between treatment arms.
Preschool and non-HEMT Pilot Cohort Safety Endpoint 5: Treatment with additional non-protocol assigned antibiotics | 28 days
  Compare treatment with additional non-protocol assigned antibiotics within the 28 days post-randomization between treatment arms.
Preschool and non-HEMT Pilot Cohort Safety Endpoint 6: Time to IV antibiotics following a randomized PEx | 28 days
  Compare time to IV antibiotics following a randomized PEx (using CF Foundation Patient Registry data, if available) between treatment arms.
Preschool and non-HEMT Pilot Cohort: Future Larger Clinical Trial Feasibility 1 | 28 days
  Measure the proportion of approached patients that enrolls.
Preschool and non-HEMT Pilot Cohort: Future Larger Clinical Trial Feasibility 2 | 28 days
  Measure the proportion of respiratory symptoms meeting randomization criteria.
Preschool and non-HEMT Pilot Cohort: Future Larger Clinical Trial Feasibility 3 | 28 days
  Measure the proportion of respiratory symptoms meeting randomization criteria resulting in treatment initiation within assigned arm.
Preschool and non-HEMT Pilot Cohort: Future Larger Clinical Trial Feasibility 4 | 28 days
  Through targeted qualitative interviews of caregivers we will describe caregivers' experience managing study treatment and report themes that emerge regarding caregivers' experiences in order to understand motivations, benefits and challenges associated with assigned treatment arm.
Clinic Throat Swab Substudy 1: Metagenomic Sequencing | 1 year
  Use quantitative polymerase chain reaction (qPCR) and metagenomic sequencing to quantitatively define throat swab microbiology at baseline, at exacerbation diagnosis, and after treatment. Metagenomic sequencing analyzes the genomes of all microorganisms in a sample, providing a broad overview of the ecosystem's composition. It can be used to study the diversity of bacteria, detect the abundance of microbes, and study unculturable microorganisms.
Clinic Throat Swab Substudy 2: Microbiota Measures | 1 year
  Correlate throat microbiota measures (both pre-treatment microbial taxonomic or functional gene abundances, and changes in those abundances) with clinical outcome measures within antibiotic treatments.
Home Throat and Nasal Swab Substudy 1: Feasibility of Home Collection of Nasal Swabs for Viral Testing and Illness Frequency | 28 days
  Assess the feasibility of home collection of nasal swabs for viral testing at the time of pulmonary exacerbation (PEx) and determine the frequency of viral illness at the time of PEx diagnosis.
Home Throat and Nasal Swab Substudy 2: Feasibility of Home Collection of Throat Swabs for Bacterial testing | 28 days
  Assess the feasibility of home collection of throat swabs for bacterial testing at the time of pulmonary exacerbation (PEx).
Home Throat and Nasal Swab Substudy 3: Association Between Viral Illness and Symptom recovery | 28 days
  Evaluate the association between the presence of viral illness and symptom recovery (number of days to recover to baseline CRISS score) between treatment arms. The Chronic Respiratory Infection Symptom Score (CRISS) ranges from 0 to 100, with higher scores indicating more symptoms.
Home Throat and Nasal Swab Substudy 3: Association Between Viral Illness and FEV1 | 28 days
  Evaluate the association between the presence of viral illness and spirometry-measured forced expiratory volume (FEV1) at Day 28.
Home Throat and Nasal Swab Substudy 3: Association Between Viral Illness and antibiotic treatment. | 28 days
  Evaluate the association between the presence of viral illness and the percent of subjects in the tailored therapy arm requiring antibiotic treatment.
Home Throat and Nasal Swab Substudy 5: Bacterial Pathogen Identification, Frequency and Impact on Treatment Changes | 28 days
  Determine the concordance of bacteria identified on CF pathogen testing at the time of pulmonary exacerbation (PEx) compared to the most recent routine clinic visit. In addition, assess how frequently new bacterial pathogens are identified at the time of PEx and how this impacts treatment changes, including the need to change or add antibiotic therapy.
Remote Monitoring Substudy 1: Feasibility of Home Spirometry Use During PEx | 28 days
  Describe the feasibility and user acceptability of home spirometry during pulmonary exacerbations (PEx) in children with CF via survey of participants at the end of the study.
Remote Monitoring Substudy 2: Feasibility of BioButton Use During PEx | 14 days
  Describe the feasibility and user acceptability of BioButton use during pulmonary exacerbations in children with CF via survey of participants at the end of the study.
Remote Monitoring Substudy 3: Change in FEV1 by Home Spirometry | 28 days
  Describe the change from nearest baseline-state FEV1 to Day 0 exacerbation state measurement and the trajectory of change during the exacerbation state (through Day 28).
Remote Monitoring Substudy 4: Compare Home Spirometry vs. Clinic Spirometry Measures | 28 days
  Compare measurements and their change measured by home spirometry vs. clinic spirometry during the exacerbation state.
Remote Monitoring Substudy 5: BioButton-measured Change in Resting Heart Rate During PEx | 14 days
  Describe changes in resting heart rate from Day 0 to 14 of the exacerbation state.
Remote Monitoring Substudy 5: BioButton-measured Change in Resting respiratory rate During PEx | 14 days
  Describe changes in Resting respiratory rate from Day 0 to 14 of the exacerbation state.
Remote Monitoring Substudy 5: BioButton-measured Change in Activity Level During PEx | 14 days
  Describe changes activity level, measured using actigraphy, and summarized as the mean (SD) number of active minutes in a day, from Day 0 to 14 of the exacerbation state.
Remote Monitoring Substudy 5: BioButton-measured Change in Sleep During PEx | 14 days
  Describe changes in sleep time from Day 0 to 14 of the exacerbation state.
Remote Monitoring Substudy 6: Compare BioButton-measured Change in resting heart rate During PEx with Baseline Averages | 14 days
  Compare changes in resting HR to averages from a 7-day period during baseline state.
Remote Monitoring Substudy 6: Compare BioButton-measured Change in Resting respiratory rate During PEx with Baseline Averages | 14 days
  Compare changes in BioButton-measured Resting respiratory rate to averages from a 7-day period during baseline state.
Remote Monitoring Substudy 6: Compare BioButton-measured Change in activity level During PEx with Baseline Averages | 14 days
  Compare BioButton-measured change in activity level during pulmonary exacerbation (PEx) to averages from a 7-day period during baseline state.
Remote Monitoring Substudy 6: Compare BioButton-measured Change in Sleep During PEx with Baseline Averages | 14 days
  Compare BioButton change in sleep during PEx to averages from a 7-day period during baseline state.
Remote Monitoring Substudy 7: Determine correlations between changes in FEV1 and CRISS to Resting Heart Rate (HR) | 14 days
  Determine correlations between changes from Day 0 to 14 in forced expiratory volume (FEV1) and CRISS score to Resting Heart Rate (HR). The Chronic Respiratory Infection Symptom Score (CRISS) ranges from 0 to 100, with higher scores indicating more symptoms.
Remote Monitoring Substudy 7: Determine correlations between changes in FEV1 and CRISS to Resting Respiratory rate | 14 days
  Determine correlations between changes from Day 0 to 14 in forced expiratory volume (FEV1) and CRISS score to Resting Respiratory rate. The Chronic Respiratory Infection Symptom Score (CRISS) ranges from 0 to 100, with higher scores indicating more symptoms.
Remote Monitoring Substudy 7: Determine correlations between changes in FEV1 and CRISS to Activity level | 14 days
  Determine correlations between changes from Day 0 to 14 in forced expiratory volume (FEV1) and CRISS score to Activity level, measured with actigraphy. The Chronic Respiratory Infection Symptom Score (CRISS) ranges from 0 to 100, with higher scores indicating more symptoms.
Remote Monitoring Substudy 7: Determine correlations between changes in FEV1 and CRISS to Sleep duration | 14 days
  Determine correlations between changes from Day 0 to 14 in forced expiratory volume (FEV1) and CRISS score to sleep duration. The Chronic Respiratory Infection Symptom Score (CRISS) ranges from 0 to 100, with higher scores indicating more symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: D. B. Sanders, MD, MS, Principal Investigator — Indiana University; Margaret Rosenfeld, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (33):
- United States (31):
  - The Children's Hospital Alabama & University of Alabama at Birmingham, Birmingham, Alabama
  - Tucson Cystic Fibrosis Center, Tucson, Arizona
  - Children's Hospital of Los Angeles & Anton Yelchin Cystic Fibrosis Clinic, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Rady Children's Hospital at University of California San Diego, San Diego, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta & Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago & Northwestern University, Chicago, Illinois
  - Riley Hospital for Children & Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Hospital, Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital & Harvard University, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The Minnesota Cystic Fibrosis Center & University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - St. Louis Children's Hospital & Washington University School of Medicine, St Louis, Missouri
  - University of Rochester Medical Center Strong Memorial, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia & University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC & University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern & Children's Health, Dallas, Texas
  - Texas Children's Hospital & Baylor College of Medicine, Houston, Texas
  - Vermont Children's Hospital & University of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Children's Wisconsin & Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children & Toronto Canada CF Centre Pediatrics, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sanders DB, Bartz TM, Zemanick ET, Hoppe JE, Hinckley Stukovsky KD, Cogen JD, Bendy L, McNamara S, Enright E, Kime NA, Kronmal RA, Edwards TC, Morgan WJ, Rosenfeld M. A Pilot Randomized Clinical Trial of Pediatric Cystic Fibrosis Pulmonary Exacerbations Treatment Strategies. Ann Am Thorac Soc. 2023 Dec;20(12):1769-1776. doi: 10.1513/AnnalsATS.202303-245OC. PMID 37683122
- See also: STOP PEDS Pilot Study manuscript — https://pubmed.ncbi.nlm.nih.gov/37683122/